CLINICAL TRIAL: NCT01657175
Title: Quality of Life and Supportive Care Needs After Oesophageal or Gastric Cancer Surgery.
Brief Title: Quality of Life After Oesophageal or Gastric Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009 /117
Record Dates: First submitted 2012-06-29; First posted 2012-08-06 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Quality of Life; Oesophageal Cancer; Gastric Cancer
Keywords: Cancer; long-term follow-up; quality of life; Surgery; Nursing
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supportive care (Experimental): The patients randomized to the supportive care arm get an extended supportive care during the first year after surgery.
  Interventions: Other: Supportive care
- Control (No Intervention): The patients randomized to the control group get "care as usual"

INTERVENTIONS:
Other: Supportive care — The patients will be randomized to control or supportive care groups.
  The control group will be given "care as usual" wich include clinical follow-ups at the surgical department.
  The supportive care group get in addition to the clinical follow-ups a supportive care programme including:
  * Discharge information about surgery and life after surgery together with their relatives.
  * Active telephone contacts 1/week th first month the 2/month up to six month after discharge by a specialized nurs.
  * Open telephone line were the patients can call the nursed ruing daytime. Discharge: approximately 2-4 weeks after surgery
  Arms: Supportive care

SUMMARY:
This study aim to assess quality of life of patients 0-5 years after oesophageal or gastric cancer surgery and to develop and test an information and support program aiming to enhance the patients quality of life (QOL) after surgery. The project contains 3 part-studies focusing on the patients life after surgery.

Data will be collected through focus group interviews and a randomized controlled trial (RCT) study.

DETAILED DESCRIPTION:
Introduction:

Patients who have undergone oesophageal resections for cancer have shown reduced quality of life (QOL) during substantial time after surgery. Postoperatively, patients are faced with extensive changes in their daily life including reduced physical and sometimes psychological capacities, problems that may be underestimated by the health care providers.

Worldwide oesophageal cancer is the 8th and gastric cancer the 4th most common cancer diagnoses (National Board of Health and Welfare, 2009). In 2009 in Sweden there were 443 new cases of oesophageal cancer and 882 of gastric cancer (total number of inhabitants in 2009, 9.4 million). Surgery, alone or in combination with chemotherapy or radiotherapy, is the only established treatment and thus offers the only possibility of a cure. After oesophagectomy or gastrectomy the planned hospital stay is approximately two to three weeks, and the expected recovery period is at least one year. The prolonged recovery period is pointed out as an energy-requiring process including physiological, psychological, social and habitual recovery, which increases the challenges for this group of patients after surgery. Even though survival after surgery, for both oesophageal and gastric cancer, has gradually improved, the 5-year survival rate remains at only 28% respectively 27%.

Aim:

The aim of this project is to assess quality of life of patients 0-5 years after oesophageal or gastric cancer surgery and to develop and test an information and support program aiming to enhance the patients QOL after surgery.

The project contains 3 part-studies that focus on the patients life after surgery.

Method:

In both studies patients that when through oesophagectomy or gastrectomy due to cancer is included. Patients that has suffered a relapse of their cancer disease, are unable to communicate in Swedish or has went through a acute surgery is not included.

Study I and II:

This studies is carried out in accordance with a descriptive explorative design focusing on I: The patients subjective experience of their QOL and II: The patients´ experience and need of supportive care, after surgery for oesophageal/gastric cancer. Data collection is carried out using semi-structured focus group interviews. A total of 17 participants divided into 4 focus groups are included (2-5 years after elective surgery) in the study. Data are to be analysed with qualitative content analysis focusing on the patients experiences of their supportive care needs after surgery.

Study III:

This study is a randomized controlled trial that focus on testing a information and support programme to patients after oesophagectomy or gastrectomy due to cancer. The intervention group gets support from a specialized nurse after surgery which contacts the patients according to a given interval during the follow up period (6 months). The control group follows the regular follow up programme that are used at the hospital where the study is conducted.

The information and support programme are evaluated through validated questionnaires that focus on quality of life (EORTC QLQ-C30 and OES-18), satisfaction whit care (EORTC INPATSAT32), sense of coherence (KASAM) and information needs (EORTC INFO 25). The patients also writes a diary regarding health care contacts after surgery.

A total number of 80 are patients are planed to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any stage tumours in the distal third of the oesophagus including type II tumours at the gastro-oesophageal junction
* Transthoracic oesophageal resection with gastric tube reconstructions and circular stapled anastomoses in the upper right chest Postoperative clinical courses without complications, and postoperative anastomotic radiograms without anastomotic leakage
* Macro and microscopically tumour free upper resection margins Willingness, physical and mental capability to comply with the result of the randomization, and ability to follow the study protocol
* Adult >18 years
* Living in the southern of Sweden (Skåne county)

Exclusion Criteria:

* Preoperative or planned postoperative chemotherapy or radiotherapy to the tumour area known at the time of discharge from the hospital.
* Postoperative need for continuous treatment with proton pump inhibitors (PPIs) or histamine-2 blockers. Treatment with steroidal or non steroidal anti inflammatory drugs other than occasionally
* Known allergy or side effects to PPIs preventing continuous treatment for one year
* Present drug or alcohol abuse
* Failure to attend at least one postoperative visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Change of QOL from discharge (discharge= approximately 2-4 weeks after surgery) to 6 months after discharge
  Quality of life will be measured at discharge, 2 weeks, 2, 4 and 6 months after discharge (discharge= approximately 2-4 weeks after surgery).
  Quality of life is evaluated using EORTC quality of life instruments at discharge and 2 weeks, 2,4 and 6 months after discharge.

SECONDARY OUTCOMES:
Satisfaction with care | At dischage, 2 weeks, 2, 4 and 6 months after discharge.
  Satisfaction with care is evaluated using EORTC satisfaction with care instruments at discharge and 2 weeks, 2,4 and 6 months after discharge.
  Discharge: approximately 2-4 weeks after surgery
Informational need | At dischage, 2 weeks, 2, 4 and 6 months after discharge.
  Informational needs is evaluated using EORTC INFO 25 instrument, at discharge and 2 weeks, 2,4 and 6 months after discharge.
  Discharge: approximately 2-4 weeks after surgery
sense of coherence (KASAM) | At dischage, 2 weeks, 2, 4 and 6 months after discharge.
  KASAM is evaluated using the KASAM instrument, at discharge and 2 weeks, 2,4 and 6 months after discharge.
  Discharge: approximately 2-4 weeks after surgery
Contacts with the health care system | At dischage, 2 weeks, 2, 4 and 6 months after discharge.
  Contacts with the health care system is evaluated through a diary at the time for the discharge and 2 weeks, 2,4 and 6 months after discharge.
  Discharge: approximately 2-4 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jan Johansson, MD PHD, Study Director — Department of surgery, Skåne university hospital
Locations (1):
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No